CLINICAL TRIAL: NCT01126034
Title: Improving Metoclopramide Prescribing Practices at Penn Through a Physician-targeted Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: UPenn - 802142
Record Dates: First submitted 2010-05-17; First posted 2010-05-19 (Estimated); Last update posted 2015-12-04 (Estimated); Status verified 2015-12

CONDITIONS: Gastroesophageal Reflux Disease; Diabetic Gastroparesis
Keywords: Metoclopramide; Randomized Controlled Trial
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- intervention (Experimental): Physicians in the intervention group were mailed a written feedback letter regarding their patients who were prescribed questionable metoclopramide therapy. Non-intervention providers received no letter. The letter consisted of the following components:
  1. The name and medical record # of the patients involved
  2. Information regarding the metoclopramide prescription: dates, dosage, indication recorded, and the duration of therapy
  3. A reminder of the adverse effect of long-term metoclopramide therapy
  4. A recommendation to consider having the patient undergo a trial of metoclopramide discontinuation if appropriate, and documentation of a discussion of risk and benefits of metoclopramide therapy with patients
  5. A request that the physician document the discontinuation trial in the electronic medical record
  Interventions: Other: intervention letter
- non-intervention (No Intervention): No intervention letters were sent to subjects in this arm

INTERVENTIONS:
Other: intervention letter — Physicians in the intervention group were mailed a written feedback letter regarding their patients who were prescribed questionable metoclopramide therapy. Non-intervention providers received no letter. The letter consisted of the following components:
  1. The name and medical record # of the patients involved
  2. Information regarding the metoclopramide prescription: dates, dosage, indication recorded, and the duration of therapy
  3. A reminder of the adverse effect of long-term metoclopramide therapy
  4. A recommendation to consider having the patient undergo a trial of metoclopramide discontinuation if appropriate, and documentation of a discussion of risk and benefits of metoclopramide therapy with patients
  5. A request that the physician document the discontinuation trial in the electronic medical record
  Arms: intervention

SUMMARY:
The investigators hypothesized that:

1) an intervention targeted at the prescribing physician would increase the rate of a metoclopramide discontinuation among patients prescribed the medication for questionable or unclear indications; and 2) the discontinuation would be durable.

ELIGIBILITY:
Inclusion Criteria:

* Physicians at University of Pennsylvania Health System who ordered an active metoclopramide prescription with a questionable indication.

Exclusion Criteria:

* Physicians-in-training (e.g., residents, fellows)
* Physicians how were investigators on this study
* Physicians serving on the the University of Pennsylvania Drug Use and Effects Committee or Information Technology Oversight Board

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2007-03; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Discontinuation of metoclopramide therapy | 12 weeks after intervention period
  Twelve weeks after the intervention period, we searched the medical records of patients in the intervention and non-intervention groups to determine whether discontinuation of metoclopramide therapy had taken place.

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Xiao Yang, MD, MSCE, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania Center for Clinical Epidemiology and Biostatistics, Philadelphia, Pennsylvania, United States